CLINICAL TRIAL: NCT02072317
Title: Paclitaxel Plus Raltitrexed Plug Compare With Taxol Second-line Treatment for Advanced Gastric Cancer Stage II Randomized Controlled Clinical Studies
Brief Title: Paclitaxel Plus Raltitrexed Plug Compare With Taxol Second-line Treatment for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, attending, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: guoweijian-2013-raltitrexed
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Advanced Gastric Cancer
Keywords: PFS
MeSH Terms: interventions — raltitrexed; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel plus raltitrexed (Experimental): taxol 135 mg/m2, raltitrexed 3 mg/m2 ivgtt d1, every three weeks for a cycle
  Interventions: Drug: taxel plus raltitrexed
- taxol (Active Comparator): taxol 135 mg/m2, every three weeks for a cycle
  Interventions: Drug: taxol

INTERVENTIONS:
Drug: taxel plus raltitrexed — taxol 135 mg/m2, raltitrexed 3 mg/m2 ivgtt d1, every three weeks for a cycle
  Arms: Paclitaxel plus raltitrexed
Drug: taxol — taxol 135 mg/m2, every three weeks for a cycle
  Arms: taxol

SUMMARY:
The purpose of this study is to evaluate and compare safety and effectiveness of Chemotherapy in Paclitaxel plus raltitrexed plug compare with taxol second-line treatment for advanced gastric cancer

DETAILED DESCRIPTION:
from the first cycle of treatment (day one) to two month after the last cycle

ELIGIBILITY:
Inclusion Criteria:

1.18~75 years old 2.Pathological diagnosis of gastric cancer or gastroesophageal junction adenocarcinoma 3.patient failed after The first line treatment of 5-Fu and platinum ,patient relapse half year after using 5 - Fu and platinum as Postoperative adjuvant chemotherapy 4.ECOG 0-1 5.At least one measurable objective tumor lesions 6.ANC≥1.5*109/L；PLT≥80*109/L；HB≥90g/L；TBI≤1.5(UNL); ALT、AST≤1.5ULN； Cr≤ULN；Ccr≥60ml/min 7.Expected survival period for 3 months or more 8. patients with voluntary participation, and sign the informed consent

Exclusion Criteria:

1. Recurrence after transfer have received taxol or docetaxel as first-line chemotherapy,If the adjuvant chemotherapy with paclitaxel,From the last chemotherapy for 6 months or less
2. With uncontrollable large pleural or peritoneal effusion
3. In the near future has a history of myocardial infarction (3 months)
4. Malignant tumour of the past five years with other organizations to source, but the full treatment of cervical carcinoma in situ and except skin basal cell carcinoma and squamous cell carcinomas;
5. With brain metastasis
6. Severe uncontrolled medical disease or acute infection
7. Pregnancy or breast-feeding women
8. Has a long history of chronic diarrhea, or now complete intestinal obstruction patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Since the date of random to disease progression or any cause of death，the average time is 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China